CLINICAL TRIAL: NCT05249660
Title: Effect of Instrument Assisted Soft Tissue Mobilization Versus Trigger Points Release on Pain; Mobility and Function of Upper Trapezius Trigger Points in Chronic Neck Pain.
Brief Title: Instrument Assisted Soft Tissue Mobilization Versus Trigger Points Release on Upper Trapezius Trigger Points
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: REC/RCR&AH/21/0129/TAUSEEF
Record Dates: First submitted 2022-02-04; First posted 2022-02-22 (Actual); Last update posted 2022-11-28 (Actual); Status verified 2022-11

CONDITIONS: Trigger Points
Keywords: Upper trapezius pain

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Soft tissue release technique (Experimental): Patient sat on a chair. The therapist stood behind the participant and held one hand over head as the support, with the thumb of the other hand scan to detect the painful area of the latent TP of the upper trapezius muscle along the fibers. Then, pressure was applied by the thumb and the participant was asked to simultaneously actively change the muscle from shorted position to elongated state (ipsilateral side flexion of the cervical to the opposite side). This technique was repeated 3-5 times per session, and each repetition was maintained for 40-60 s till release is felt, with a 15-second rest interval. Three times passive stretching of the upper trapezius muscle was also performed for 45 s for each side.
  Interventions: Other: Soft tissue release technique
- Instrument assisted soft tissue mobilization (Active Comparator): Patient lied prone; the treatment was applied for approximately 20-seconds in a direction parallel to the muscle fibers with the instrument at a 45º angle. Followed immediately by treating the muscles in a direction perpendicular to the muscle fibers with the instrument at a 45º angle for an additional 20-second, resulting in a total treatment time of approximately 40 s. This technique was applied 3-5 times per session with 20 s rest between each time. Three times passive stretching of the upper trapezius muscle was also performed for 45 s for each side.
  Interventions: Other: Comparator: Instrument assisted soft tissue mobilization

INTERVENTIONS:
Other: Soft tissue release technique — Patient sat on a chair. The therapist stood behind the participant and held one hand over head as the support, with the thumb of the other hand scan to detect the painful area of the latent TP of the upper trapezius muscle along the fibers. Then, pressure was applied by the thumb and the participant was asked to simultaneously actively change the muscle from shorted position to elongated state (ipsilateral side flexion of the cervical to the opposite side). This technique was repeated 3-5 times per session, and each repetition was maintained for 40-60 s till release is felt, with a 15-second rest interval. Three times passive stretching of the upper trapezius muscle was also performed for 45 s for each side.
  Arms: Soft tissue release technique
Other: Comparator: Instrument assisted soft tissue mobilization — Patient lied prone; the treatment was applied for approximately 20-seconds in a direction parallel to the muscle fibers with the instrument at a 45º angle. Followed immediately by treating the muscles in a direction perpendicular to the muscle fibers with the instrument at a 45º angle for an additional 20-second, resulting in a total treatment time of approximately 40 s. This technique was applied 3-5 times per session with 20 s rest between each time. Three times passive stretching of the upper trapezius muscle was also performed for 45 s for each side.
  Arms: Instrument assisted soft tissue mobilization

SUMMARY:
Study will be randomized clinical trial. Data will be collected from non probability consecutive sampling technique. Total 30 participants from Ganga Ram Hospital and Care medical centre will be selected and randomly allocated to two different groups i.e Group A and Group B. . Group A will be treated by trigger point release. Group B will be treated by Instrument assisted soft tissue release. NPRS, GONIOMETRY, NDI will be used as outcome measuring tool before and after treatment. Data will be analyzed by using Statistical package for social sciences 25.

DETAILED DESCRIPTION:
Trigger point is defined as a hyperirritable palpable nodule contained in the skeletal muscle fibers. The palpable nodule, also named taut band, is described as a limited number of fibers with an increased stiffness. Trp causes the muscles to week and stiff, leading to reduction in range of movement. MTrP can produce local and referred pain, either on manual compression or spontaneously.

Instrument-assisted soft tissue mobilization (IASTM) is the use of hard tools to manipulate soft tissue and was derived from the Cyriax1 cross-friction massage. It has recently emerged as a popular alternative to traditional manual therapy techniques. Modern-day IASTM instruments vary in material (e.g. stainless steel, plastic) and design and are used to improve a variety of musculoskeletal conditions and associated outcomes.

Manual technique that uses direct vertical pressure to the TP, is a well-established treatment method used to resolve the TP-related pain syndrome. This directed pressure is managed according to the therapist's perception of the tissue resistance of the treated soft tissue or according to the pain perceived by the patient based on a pain scale. Manual therapy is a commonly used treatment for MPS as it has been considered one of the most effective techniques for the inactivation of MTrPs.

ELIGIBILITY:
Inclusion Criteria:

* Patients with neck pain in the upper trapezius muscle
* Tender nodule, constant pain, a jump sign during palpation will be included in this study

Exclusion Criteria:

* Patients with Whiplash injury
* History of neck/shoulder surgery
* Cervical Radiculopathy
* History of malignancy

Ages: 20 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30 (Actual)
Dates: Start 2022-01-25 (Actual); Primary Completion 2022-07-13 (Actual); Study Completion 2022-07-13 (Actual)

PRIMARY OUTCOMES:
Numeric pain rating scale | 6 weeks
  Scale consists of 4 questions regarding actual pain level, zero indicates no pain and 10 indicates worst pain imaginable
Goniometry | 6 weeks
  Goniometer is used to measure the ranges of body joints.
Neck disability index | 6 weks
  Scale consists of 10 sections,each section contains questions regarding head/ neck pain and some questions regarding the daily activities that we perform

CONTACTS AND LOCATIONS:
Overall Officials: Muhammad Sanaullah, MS, Principal Investigator — Riphah International University
Locations (1):
- Ganga Ram Hospital and Care medical centre, Lahore, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No